CLINICAL TRIAL: NCT05413837
Title: Imaging Research on Anatomical Variation of Cerebral Venous Sinus in Healthy Individuals
Brief Title: Anatomical Variation of Cerebral Venous Sinus in Healthy Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Other Study IDs: CVSAV-HI
Record Dates: First submitted 2022-06-06; First posted 2022-06-10 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Venous Sinus Thrombosis, Cranial
Keywords: venous sinus; anatomy
MeSH Terms: conditions — Sinus Thrombosis, Intracranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples from enrolled participants are drawn by nurse using containing coagulant tubes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: anotomy and variation of venous sinus — Contrast enhanced-magnatic resonance venography（CE-MRV）and other magnetic resonance imaging methods are used to estimate the anatomy of cerebral venous sinus.
Diagnostic Test: the level of biomarker in bood — Elisa or omics analysis is used to test the level of biomarker in blood.

SUMMARY:
The anatomical characteristics of veins and venous sinus result in great differences between cerebral venous system diseases and cerebral artery diseases in etiology, pathophysiology and clinical features.Therefore, understanding the anatomy and variation of normal venous sinuses is essential to identify the intracranial venous lesions.

DETAILED DESCRIPTION:
The classification of venous sinus and its variation based on the autopsy of patients can not fully reflect the real anatomy and variation of venous sinus in human, and the targeted research on healthy people is still unknown. The main purpose of this research is to use multimodal magnetic resonance technology to study the variation of venous sinus in Chinese healthy population, to preliminarily improve the anatomical classification of venous sinus in Chinese , to verify the the correlation between venous sinus variation and various non-genetic factors at the same time, as well as establishing reliable quantitative evaluation indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 35 years old.
2. Confirmed no intracranial diseases, congenital abnormalities such as intracranial hematoma, tumor, vascular malformation, hydrocephalus, etc.
3. Voluntarily signed informed consent.

Exclusion Criteria:

1. Any clinical history, including hypertension, diabetes, coronary heart disease, hematologic and rheumatic immune system diseases,cervical spondylosis, anxiety, depression, insomnia, etc.
2. Internal jugular venous outflow disturbance : MRV from extracranial to aortic arch demonstrates variation or stenosis of the internal jugular vein, vertebral plexus, brachiocephalic vein, and superior vena cava.
3. Any history of craniocerebral trauma or surgery that affected the existence and running of veins.Unhealthy habits such as smoking, heavy drinking, etc.
4. Women who are pregnant or in preparation for pregnancy or lactation.
5. Other conditions that the researchers considered might affect the trial and inappropriate for inclusion.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Chinese healthy individuals aged 18-35 years without clinical symtoms and cerebral venous diseases
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
The anotomy and variation of venous sinus in Chinese healthy individuals | On the day of examination
  According to the connection types of superior sagittal sinus and transverse sinus at the the torcular Herophili assessed with contrast-enhanced MR venography and phase-contrast MR venography, describe the anatomical classification of venous sinus based on the anatomical descriptions of Osborn and describe the anatomical variations that are not included in the existing classification. Calculating the proportion of each type.

SECONDARY OUTCOMES:
The diameters of venous sinus and small veins in Chinese healthy individuals | On the day of examination
  Measuring the diameters of venous sinus and small veins assessed with contrast-enhanced MR venography
Serum biomarkers in Chinese healthy individuals | On the day of examination
  The level of biomarkers are detected using Elisa or omics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD.PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital;Capital Medical University, Beijin, XI Cheng District, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng Y, Li WA, Fan X, Li X, Chen J, Wu Y, Meng R, Ji X. Normal anatomy and variations in the confluence of sinuses using digital subtraction angiography. Neurol Res. 2017 Jun;39(6):509-515. doi: 10.1080/01616412.2017.1323383. Epub 2017 May 11. PMID 28494642